CLINICAL TRIAL: NCT03109821
Title: Home-based Rehabilitation Following a Total Hip Replacement - do Patients Follow the Exercise Prescription and How Does it Relate to Postoperative Recovery? The Pragmatic Home-Based Exercise After Total Hip Arthroplasty Silkeborg 1 (PHETHAS-1) Trial
Brief Title: Home-based Rehabilitation Following a Total Hip Replacement
Acronym: PHETHAS-1
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 654894
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2019-03

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Exercise Therapy; Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- THA patients
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Home-based exercise — The intervention reflects the standard rehabilitation practice at Elective Surgery Centre. 3 weeks after surgery the patients will receive a thorough instruction and supervision in the strength training exercises that they are to perform without supervision at their own homes the following 7 weeks. The instruction is conducted one-to-one by physiotherapists and supported by an instruction booklet with written and illustrated exercise descriptions. The exercises included are: hip abduction, flexion and extension with elastic band resistance and sit-to-stand and one-legged stance. The prescribed training load will be two sets with repetitions to failure and a relative load of 10 to 20 RM (Repetition Maximum), performed every second day (3-4 times a week).
  Exposure: Performed exercise dose will be quantified as the total physiological exercise stimulus (Time under tension summary dose) recorded by a sensor (BandCizer) attached to the elastic exercise band.

SUMMARY:
In this study we will investigate the relation between performed exercise dose and recovery after total hip replacement (THA). A dose-response relationship is hypothesized.

It is the primary objective to indicate the preliminary efficacy of home-based rehabilitation using elastic band exercise on performance-based function after THA, based on the relationship between the performed exercise dose (objectively quantified time under tension summary dose) and the change in 40 meter maximal gait speed (performance-based function) from 3 (start of intervention) to 10 weeks (end of intervention) after surgery.

DETAILED DESCRIPTION:
The study is a pragmatic, single center, prospective cohort study (single cohort) to be conducted in Silkeborg, Denmark. The outcomes will be collected in the period from 3 to 10 weeks after surgery by an assessor blinded to exercise compliance. The study will adhere methodologically to the STROBE guidelines and checklist for prospective cohort studies (www.strobe-statement.org).

The study design and completion is conducted in a research collaboration between the Interdisciplinary Research Unit at Elective Surgery Centre based at Silkeborg Regional Hospital and Physical Medicine & Rehabilitation Research - Copenhagen (PMR-C) based at Hvidovre Hospital.

Primary objective, eligibility criteria, exposure/intervention and outcome measures are entered elsewhere. At June 28, 2017, two outcome measures were added to the study. At 10 weeks after surgery, patients will be asked both to describe change in hip problems (from preoperatively to 10 weeks after surgery) and to describe their perception of outcome after surgery. The outcome measures will be used for exploratory analysis of patient acceptable symptom state (PASS) and minimal clinically important improvement (MCII)

Primary analysis:

A simple linear regression analysis will be performed to evaluate the association between performed exercise dose and change in score on gait speed. Furthermore descriptive statistics will be used to quantify exercise compliance and to indicate the exercise dosage with the greatest response. Patients will be divided into four compliance-quartiles and summary statistics of the primary outcome (change in gait speed) will be presented graphically to illustrate possible dose-response relationship.

Secondary analyses:

For change in patient-reported function the analysis will be similar to the analysis for change in gait speed. Summary statistics on the rest of the secondary outcomes will be presented for the compliance-quartiles.

In a multiple regression analysis the association between gait speed (at 10 weeks follow up) and self-efficacy, 24-hour physical activity, performed exercise dose and gait speed (at baseline) will be analyzed.

Furthermore summary statistics will be presented for demographic data and other pre-specified outcomes.

Additionally, an embedded qualitative study will be performed to explore motivation and barriers related to exercise compliance. This study will be reported in a secondary paper with a clear reference to the primary trial and trial registration.

Regional Hospital Central Jutland and The Danish Rheumatism Association is partly funding the salary for physiotherapists involved in the study. Further external funding will be applied for.

ELIGIBILITY:
Inclusion criteria:

* Above 18 years
* Scheduled for a primary THA, at Elective Surgery Centre, due to osteoarthritis
* Able to understand written and spoken Danish

Exclusion criteria:

* Referral to supervised rehabilitation in the municipality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage hip osteoarthritis, who are scheduled for primary THA at the Elective Surgery Centre at the public hospital, Silkeborg Regional Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | Change from 3 to 10 weeks after surgery.
  Measured by the 40m fast-paced walk test (continous, m/sec)

SECONDARY OUTCOMES:
Gait speed | 10 weeks after surgery
  Measured by the 40m fast-paced walk test (continous, m/sec)
Change in patient-reported function | Change from 3 to 10 weeks after surgery.
  Measured by the ADL (Activities of Daily Living) subscale of Hip disability and Osteoarthritis Outcome Score (HOOS). HOOS is a disease-specific patient-reported outcome measure (continous)
Change in patient-reported symptoms | Change from 3 to 10 weeks after surgery.
  Measured by the symptoms subscale of HOOS (continous)
Change in patient-reported pain | Change from 3 to 10 weeks after surgery.
  Measured by the pain subscale of HOOS (continous)
Change in patient-reported hip related quality of life | Change from 3 to 10 weeks after surgery.
  Measured by the quality of life subscale (QoL) of HOOS (continous)
Change in lower-extremity function | Change from 3 to 10 weeks after surgery
  Measured by the Chair stand test (The maximal number of rises from a chair within 30 seconds) (continous)
Change in hip abductor muscle strength | Change from 3 to 10 weeks after surgery
  Test of isometric muscle strength in hip abduction in the operated leg. The hand-held dynamometer Power Track II Commander will be used to assess this using standardized test procedures (continous, Nm/kg)
Change in hip flexor muscle strength | Change from 3 to 10 weeks after surgery
  Test of isometric muscle strength in hip flexion in the operated leg. The hand-held dynamometer Power Track II Commander will be used to assess this using standardized test procedures (continous, Nm/kg)
Self-efficacy | 3 weeks after surgery
  The general self-efficacy scale will be used to measure self-efficacy, defined as an individual's belief in his or her capacity to execute behaviors necessary to produce specific performance attainments (continous)
24-hour physical activity (mean upright time). | 4 weeks after surgery
  An ActivPAL movement-sensor will be used to measure mean time per day in upright position (standing and walking) based on 7 days of data collection. The sensor will be applied 3 weeks after surgery and used the following week (continous, min/day)
24-hour physical activity (mean number of steps) | 4 weeks after surgery
  An ActivPAL movement-sensor will be used to measure mean number of steps per day based on 7 days of data collection. The sensor will be applied 3 weeks after surgery and used the following week (continous, min/day)

OTHER OUTCOMES:
Number of participants with adverse events | 3 weeks after surgery
  Number and type of adverse events will be registered by the physiotherapist (categorical)
Number of participants with adverse events | 10 weeks after surgery
  Number and type of adverse events will be registered by the physiotherapist (categorical)
Mean change in pain after each exercise session | 10 weeks after surgery.
  The Visual Analogue Scale (VAS) will be used to assess pain before and after each exercise session. Data will be summarized as a mean change in pain per exercise session for the entire intervention period (continous)
Motivation to perform the prescribed exercises | 3 weeks after surgery
  The participants will be asked about their motivation to perform the prescribed exercises. A short questionnaire developed for this purpose will be used. The possible responses are ordered in 4 levels of motivation on a ordinal scale (categorical)

CONTACTS AND LOCATIONS:
Overall Officials: Lone R Mikkelsen, PhD, Principal Investigator — Silkeborg Regional Hospital
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Madsen MN, Mikkelsen LR, Rathleff MS, Thorborg K, Kallemose T, Bandholm T. Hip strengthening exercise dosage is not associated with clinical improvements after total hip arthroplasty - a prospective cohort study (the PHETHAS-1 study). BMC Musculoskelet Disord. 2024 Nov 19;25(1):928. doi: 10.1186/s12891-024-08057-x. PMID 39563311
- [Derived] Mikkelsen LR, Madsen MN, Rathleff MS, Thorborg K, Rossen CB, Kallemose T, Bandholm T. Pragmatic Home-Based Exercise after Total Hip Arthroplasty - Silkeborg: Protocol for a prospective cohort study (PHETHAS-1). F1000Res. 2019 Jun 25;8:965. doi: 10.12688/f1000research.19570.2. eCollection 2019. PMID 31448107